CLINICAL TRIAL: NCT06416150
Title: Reducing Urban Cervical Cancer Disparities Using a Tailored MHealth Intervention to Enhance Colposcopy Attendance
Brief Title: Reducing Urban Cervical Cancer Disparities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Rutgers, The State University of New Jersey (Other); Thomas Jefferson University (Other); Temple University (Other); University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 23-1035
Record Dates: First submitted 2024-04-09; First posted 2024-05-16 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Cervical Cancer; Papilloma Viral Infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (13):
- Stage 1 and 3 SoC (Experimental): Start with Stage 1 Standard of Care; patient attends baseline colposcopy appointment, no Stage 2 intervention. Continue with Stage 3 Standard of Care; patient attends 12-month follow-up appointment, no Stage 4 intervention.
  Interventions: Behavioral: Stage 1 SOC; Behavioral: Stage 3 SOC
- Stage 1 and 3 SoC + Stage 4 HERS (Experimental): Start with Stage 1 Standard of Care; patient attends baseline colposcopy appointment, no Stage 2 intervention. Continue with Stage 3 Standard of Care; patient does not attend 12-month follow-up appointment, continue with Stage 4 HERS intervention.
  Interventions: Behavioral: Stage 1 SOC; Behavioral: Stage 3 SOC; Behavioral: Stage 4 HERS
- Stage 1 SoC + Stage 2 and 3 HERS (Experimental): Start with Stage 1 Standard of Care; patient does not attend baseline colposcopy appointment, continue with Stage 2 HERS intervention. Continue with Stage 3 HERS intervention; patient attends 12-month follow-up appointment, no Stage 4 intervention.
  Interventions: Behavioral: Stage 1 SOC; Behavioral: Stage 2 HERS; Behavioral: Stage 3 HERS
- Stage 1 SoC + Stage 2, 3, and 4 HERS (Experimental): Start with Stage 1 Standard of Care; patient does not attend baseline colposcopy appointment, continue with Stage 2 HERS intervention. Continue with Stage 3 HERS intervention; patient does not attend 12-month follow-up appointment, continue with Stage 4 HERS intervention.
  Interventions: Behavioral: Stage 1 SOC; Behavioral: Stage 2 HERS; Behavioral: Stage 3 HERS; Behavioral: Stage 4 HERS
- Stage 1 SoC + Stage 2 and 3 HERS + Stage 4 HERS+HC (Experimental): Start with Stage 1 Standard of Care; patient does not attend baseline colposcopy appointment, continue with Stage 2 HERS intervention. Continue with Stage 3 HERS intervention; patient does not attend 12-month follow-up appointment, continue with Stage 4 HERS+HC intervention.
  Interventions: Behavioral: Stage 1 SOC; Behavioral: Stage 2 HERS; Behavioral: Stage 3 HERS; Behavioral: Stage 4 HERS+HC
- Stage 1 and 3 HERS (Experimental): Start with Stage 1 HERS intervention; patient attends baseline colposcopy appointment, no Stage 2 intervention. Continue with Stage 3 HERS intervention; patient attends 12-month follow-up appointment, no Stage 4 intervention.
  Interventions: Behavioral: Stage 1 HERS; Behavioral: Stage 3 HERS
- Stage 1, 3, and 4 HERS (Experimental): Start with Stage 1 HERS intervention; patient attends baseline colposcopy appointment, no Stage 2 intervention. Continue with Stage 3 HERS intervention; patient does not attend 12-month follow-up appointment, continue with Stage 4 HERS intervention.
  Interventions: Behavioral: Stage 1 HERS; Behavioral: Stage 3 HERS; Behavioral: Stage 4 HERS
- Stage 1 and 3 HERS + Stage 4 HERS+HC (Experimental): Start with Stage 1 HERS intervention; patient attends baseline colposcopy appointment, no Stage 2 intervention. Continue with Stage 3 HERS intervention; patient does not attend 12-month follow-up appointment, continue with Stage 4 HERS+HC intervention.
  Interventions: Behavioral: Stage 1 HERS; Behavioral: Stage 3 HERS; Behavioral: Stage 4 HERS+HC
- Stage 1, 2, and 3 HERS (Experimental): Start with Stage 1 HERS intervention; patient does not attend baseline colposcopy appointment, continue with Stage 2 HERS intervention. Continue with Stage 3 HERS intervention; patient attends 12-month follow-up appointment, no Stage 4 intervention.
  Interventions: Behavioral: Stage 1 HERS; Behavioral: Stage 2 HERS; Behavioral: Stage 3 HERS
- Stage 1, 2, 3, and 4 HERS (Experimental): Start with Stage 1 HERS intervention; patient does not attend baseline colposcopy appointment, continue with Stage 2 HERS intervention. Continue with Stage 3 HERS intervention; patient does not attend 12-month follow-up appointment, continue with Stage 4 HERS intervention.
  Interventions: Behavioral: Stage 1 HERS; Behavioral: Stage 2 HERS; Behavioral: Stage 3 HERS; Behavioral: Stage 4 HERS
- Stage, 2, and 3 HERS + Stage 4 HERS+HC (Experimental): Start with Stage 1 HERS intervention; patient does not attend baseline colposcopy appointment, continue with Stage 2 HERS intervention. Continue with Stage 3 HERS intervention; patient does not attend 12-month follow-up appointment, continue with Stage 4 HERS+HC intervention.
  Interventions: Behavioral: Stage 1 HERS; Behavioral: Stage 2 HERS; Behavioral: Stage 3 HERS; Behavioral: Stage 4 HERS+HC
- Stage 1 HERS + Stage 2 and 3 HERS+HC (Experimental): Start with Stage 1 HERS intervention, patient does not attend baseline colposcopy appointment, continue with Stage 2 HERS+HC intervention. Continue with Stage 3 HERS+HC intervention; patient attends 12-month follow-up appointment, no Stage 4 intervention.
  Interventions: Behavioral: Stage 1 HERS; Behavioral: Stage 2 HERS+HC; Behavioral: Stage 3 HERS+HC
- Stage 1 HERS + Stage 2, 3, and 4 HERS+HC (Experimental): Start with Stage 1 HERS intervention, patient does not attend baseline colposcopy appointment, continue with Stage 2 HERS+HC intervention. Continue with Stage 3 HERS+HC intervention; patient does not attend 12-month follow-up appointment, continue with Stage 4 HERS+HC intervention.
  Interventions: Behavioral: Stage 1 HERS; Behavioral: Stage 2 HERS+HC; Behavioral: Stage 3 HERS+HC; Behavioral: Stage 4 HERS+HC

INTERVENTIONS:
Behavioral: Stage 1 SOC — Participants will receive high Standard Care, consisting of a telephone call approximately one month before the appointment to confirm the appointment date for the baseline colposcopy appointment, followed by a notification letter including scheduled appointment date and clinic contact information should the clinic be unable to reach the patient by telephone.
  Arms: Stage 1 SoC + Stage 2 and 3 HERS; Stage 1 SoC + Stage 2 and 3 HERS + Stage 4 HERS+HC; Stage 1 SoC + Stage 2, 3, and 4 HERS; Stage 1 and 3 SoC; Stage 1 and 3 SoC + Stage 4 HERS
Behavioral: Stage 1 HERS — Participants will receive text message appointment reminders and barriers messages. Text messages will be sent on a prescheduled basis over the course of 2 weeks preceding the scheduled target appointment.
  Arms: Stage 1 HERS + Stage 2 and 3 HERS+HC; Stage 1 HERS + Stage 2, 3, and 4 HERS+HC; Stage 1 and 3 HERS; Stage 1 and 3 HERS + Stage 4 HERS+HC; Stage 1, 2, 3, and 4 HERS; Stage 1, 2, and 3 HERS; Stage 1, 3, and 4 HERS; Stage, 2, and 3 HERS + Stage 4 HERS+HC
Behavioral: Stage 2 HERS — Participants will receive another barriers assessment and another round of text message appointment reminders and barriers messages.
  Arms: Stage 1 SoC + Stage 2 and 3 HERS; Stage 1 SoC + Stage 2 and 3 HERS + Stage 4 HERS+HC; Stage 1 SoC + Stage 2, 3, and 4 HERS; Stage 1, 2, 3, and 4 HERS; Stage 1, 2, and 3 HERS; Stage, 2, and 3 HERS + Stage 4 HERS+HC
Behavioral: Stage 2 HERS+HC — Participants will receive another barriers assessment and another round of text message barriers counseling as well as health coaching (HC) after their missed appointment. Participants that miss their scheduled appointment will receive a HC call within 2 business days. HC calls will be flexibly scheduled based on the preference of the patients and limited to 15 minutes or less.
  Arms: Stage 1 HERS + Stage 2 and 3 HERS+HC; Stage 1 HERS + Stage 2, 3, and 4 HERS+HC
Behavioral: Stage 3 SOC — Participants will receive a telephone call before their 12-month follow-up appointments to remind participants about their upcoming appointment and schedule/reschedule if needed.
  Arms: Stage 1 and 3 SoC; Stage 1 and 3 SoC + Stage 4 HERS
Behavioral: Stage 3 HERS — Participants will receive text message appointment reminders and barriers messages. Text messages will be sent on a prescheduled basis over the course of 2 weeks preceding the scheduled target appointment.
  Arms: Stage 1 SoC + Stage 2 and 3 HERS; Stage 1 SoC + Stage 2 and 3 HERS + Stage 4 HERS+HC; Stage 1 SoC + Stage 2, 3, and 4 HERS; Stage 1 and 3 HERS; Stage 1 and 3 HERS + Stage 4 HERS+HC; Stage 1, 2, 3, and 4 HERS; Stage 1, 2, and 3 HERS; Stage 1, 3, and 4 HERS; Stage, 2, and 3 HERS + Stage 4 HERS+HC
Behavioral: Stage 3 HERS+HC — Participants will receive text message barriers counseling as well as HC after their missed appointment. Participants that miss their scheduled appointment will receive a HC call within 2 business days. HC calls will be flexibly scheduled based on the preference of the patients and limited to 15 minutes or less.
  Arms: Stage 1 HERS + Stage 2 and 3 HERS+HC; Stage 1 HERS + Stage 2, 3, and 4 HERS+HC
Behavioral: Stage 4 HERS — Participants will receive another barriers assessment and another round of text message appointment reminders and barriers messages.
  Arms: Stage 1 SoC + Stage 2, 3, and 4 HERS; Stage 1 and 3 SoC + Stage 4 HERS; Stage 1, 2, 3, and 4 HERS; Stage 1, 3, and 4 HERS
Behavioral: Stage 4 HERS+HC — Participants will receive another barriers assessment and another round of text message barriers counseling as well as HC. Participants that miss their scheduled appointment will receive a HC call within 2 business days. HC calls will be flexibly scheduled based on the preference of the patients and limited to 15 minutes or less.
  Arms: Stage 1 HERS + Stage 2, 3, and 4 HERS+HC; Stage 1 SoC + Stage 2 and 3 HERS + Stage 4 HERS+HC; Stage 1 and 3 HERS + Stage 4 HERS+HC; Stage, 2, and 3 HERS + Stage 4 HERS+HC

SUMMARY:
This study uses a hybrid Type 1 effectiveness-implementation trial to operationalize and assess the efficacy of the Health Enhancement Resource System (HERS) intervention. HERS aims to increase patient follow-up after abnormal test results through text message-based barriers counseling for women and supplemental telephone-based Health Coaching for women who miss their appointment.

DETAILED DESCRIPTION:
Invasive cervical cancer is preventable with well-established screening and diagnostic tests. However, there is a large and persistent disparity gap in cervical cancer mortality rates among urban, underserved populations that continues to intensify. This gap is largely due to low follow-up after an abnormal test result leading to continued disease risk.

The study team developed an efficacious, tailored telephone counseling intervention delivered by a health coach [Tailored Communication for Cervical Cancer Risk (TC3)] that increased attendance at follow-up appointments for initial colposcopy among urban, underserved women. This evidence-based intervention is available for dissemination and implementation through the National Cancer Institute's Evidence-based Cancer Control Programs database. However, TC3 was developed prior to the upsurge of smartphones and texting usage and is resource-intensive, requiring dedicated staff to interview and counsel patients before their appointment, limiting its scalability and sustainability. Therefore, this study proposes use of a hybrid type 1 effectiveness-implementation study design to assess the impact of a Health Enhancement Resource System (HERS)-adapted from TC3-on attending follow-up appointments after an abnormal cervical test result.

Using a sequential, multiple assignment, randomized trial (SMART) design, a multi-site intervention study will be conducted at three high-volume, urban clinic sites in PA and NJ serving predominately low-income minority women: Fox Chase Cancer Center/Temple University Health System; Rutgers University, and Thomas Jefferson University. The study will target patients scheduled for first time or repeat colposcopy through (a) HERS text message-based barriers counseling and (b) supplemental telephone-based Health Coaching for women who miss their scheduled appointment.

Participants scheduled for a colposcopy after an abnormal cervical test will be recruited and randomized in a 1:1 ratio to receive either Standard of Care or HERS (text message intervention). Participants randomized to Standard of Care who do not attend the scheduled colposcopy appointment will be assigned to receive HERS. Participants randomized to HERS who do not attend the scheduled colposcopy appointment will be rerandomized to receive either HERS (repeating the text message intervention) or HERS+HC (text plus health coaching).

For the 12-month colposcopy appointment, participants will continue with the last intervention assignment they completed for the first colposcopy appointment (i.e., Standard of Care, HERS, or HERS+HC). Again, participants randomized to Standard of Care who do not attend the 12-month scheduled colposcopy appointment will be assigned to receive HERS. Participants randomized to HERS who do not attend the 12-month scheduled colposcopy appointment will be rerandomized to receive either HERS (repeating the text message intervention) or HERS+HC (text plus health coaching). Participants randomized to HERS+HC who do not attend the 12-month scheduled colposcopy appointment will be assigned to repeat HERS+HC.

All participants will complete surveys at baseline survey and a 1-week post-appointment survey for both colposcopy appointments. Participants will also complete a barriers assessment. Standard of Care participants will complete the assessment via online survey while HERS and HERS+HC participants will complete the barriers assessment via text message as part of the HERS text message intervention.

Qualitative interviews will be completed with providers at each site at pre-implementation and post-implementation. Additionally, a subset of participants will complete exit interviews after their 12-month colposcopy appointment.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 90 years of age (screening is still recommended for some women over 65-depending on screening and medical history and proceeds until age 90 in the study's clinic recruitment sites),
* referral for colposcopic evaluation at the clinic sites,
* able to communicate with ease in English,
* have a cell phone with texting ability, and
* competent to give consent.

Exclusion Criteria:

* are pregnant at the time of recruitment,
* display current evidence or have a history of positive invasive carcinoma of the cervix, or
* require follow-up but not a colposcopy.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 546 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Attendance at baseline colposcopy appointment | Up to 3 months post-baseline
  Patient attendance or non-attendance at baseline colposcopy appointment assessed via appointment attendance history in electronic medical records

SECONDARY OUTCOMES:
Attendance at 12-month follow-up appointment | Up to 15 months post-baseline
  Patient attendance or non-attendance at 12-month follow-up appointment assessed via appointment attendance history in electronic medical records

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne M Miller, PhD, Principal Investigator — Fox Chase Cancer Center
Locations (3):
- United States (3):
  - Rutgers, The State University of New Jersey, New Brunswick, New Jersey
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data sharing is essential to increase reproducibility and transparency of research and the translation of research findings into practice, leading to improved health outcomes. Data generated from the proposed study will be shared with the research community through presentations at scientific meetings and publications in peer-reviewed journals. Further, data will be available to qualified researchers after the main findings are published in a peer-reviewed journal. All data sharing will comply with local, state, and federal laws and regulations, including HIPAA Privacy and Security Rules. Data will be de-identified before presentations and publications, as well as any datasets shared with qualified researchers.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Study data will be available after publication of the main study outcomes.
Access Criteria: Contact the study PI to request data or supporting information.
URL: http://www.foxchase.org/suzanne-miller